CLINICAL TRIAL: NCT05222763
Title: Effect Of Web - Supported Interactıve Nursıng Program After Mastectomy On Body Value, Care Dependence And Psychosocıal Adaptatıon To Dısease-Self-Awareness Levels Accordıng To Self-Regulatıon Model: Mıxed Method Study
Brief Title: Web-Assisted Interactive Nurse Program in Mastectomy Patients: A Mixed Method Study
Acronym: Mastectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cumhuriyet University (Other)
Responsible Party: Principal Investigator, Şeyda KAZANÇ, Lecturer, Cumhuriyet University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 939597
Record Dates: First submitted 2022-01-24; First posted 2022-02-03 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Web Based Intervention; Mastectomy; Illness Perception; Nursing Caries
Keywords: Mastectomy; body value; adaptation to illness; care addiction

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients participating in the study will know that they are in a randomized controlled study, but they will not know which group they are in until the study is completed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Interventional group (Experimental): The web-supported interactive nursing program intervention will take 3 weeks. The first week of the training will begin with the patient's admission to the clinic. Shoulder and Arm Exercises, Lymphedema in the Arm and Prevention of Its Development, and qualitative study, the themes of misperception determined in this area will be emphasized. In the second week, they will be asked to continue their Shoulder and Arm Exercises training, to examine the Other Side Breast Examination Training and Adaptation Process to Life Activities, Skin Care and Post-Surgery Cancer Treatment and Breast Reconstruction. In the last week of the training, it will be requested to review the contents again. Correct perceptions that may emerge as a result of the qualitative study will be supported in the relevant parts of the training. During the study, short mobile phone messages containing reminders and motivations will be sent regularly twice a week (8 times).
  Interventions: Behavioral: Web-assisted patient education intervention designed according to the self-regulation model
- Behavioral: (Active Comparator): The handbook developed within the scope of the "Women's Return to Social Life After Mastectomy" Project on the website of the Continuing Education, Research and Solidarity Association will be used on the website of the participants assigned to the control group.
  Interventions: Behavioral: The website where the mastectomy patients handbook

INTERVENTIONS:
Behavioral: Web-assisted patient education intervention designed according to the self-regulation model — Implementation of patient education with the website created about care and compliance needs in mastectomy patients obtained as a result of qualitative research.
  Arms: Experimental: Interventional group
Behavioral: The website where the mastectomy patients handbook — The site where the patient booklet is available as pdf
  Arms: Behavioral:

SUMMARY:
This study is planned to examine the levels of bodily value, care dependence and psychosocial cohesion-self-notification of patients in the Web Assisted Interactive Nursing Program (WDIHP) designed according to the Self Regulation Model. The mixed method is a research. One of the mixed research methods, the discovery sequenced design, will be used. The research will continue with the quantitative part, starting with the qualitative part. The quantitative part of the research is a randomized controlled experimental trial.

DETAILED DESCRIPTION:
Complications after surgery are common in patients who undergo mastectomies, as in every surgery. Mastectomy patients need to protect the wound area and the arm on the side where a mastectomy is performed following surgery. The process of wound healing and return to the patient's daily life in the post-surgery process parallels. In the early post-operative period, patients have difficulty carrying out daily living activities and need support, while in the late-term they are able to perform daily living activities more independently from caregivers and nurses.

Objective: This research was planned to examine the body value of mastectomy patients, care dependence and psychosocial adaptation-self-knowledge levels of the Web Assisted Interactive Nursing Program (WDIHP) designed according to the Self-Regulation Model.

Method: The research is designed as a mixed-method study of qualitative-quantitative research methods, designed according to the Self-Regulation Model, to examine the effect of WDHP on adaptation to social life, self-efficacy, and body value in patients undergoing breast cancer surgery. This study will use exploratory hybrid methods from mixed research methods. Qualitative interviews will be held face-to-face. Interviews with participants will continue until data saturation is achieved. In the qualitative part of the research, the in-depth interview method will be selected and the "Semi-Structured Interview Form" will be used as a data collection tool. All interviews will be recorded in digital format, returned to writing and then transferred to qualitative analysis software MAXQDA. The quantitative part of the study will be carried out as a randomized controlled trial using the block randomization method. Randomization will be done by a statistician other than the researcher. Power analysis was calculated using G * Power 3.1.9.7 program. With 0.95 effect size, 95% power and 0.05 significance level, the required sample size was determined as 30 individuals per group, and 60 individuals in total. It was decided to include 67 individuals, 35 individuals in the intervention group and 31 individuals in the control group, by taking 15% more of the calculated sample against the possibility of sample loss during the study. The correct perceptions that may arise as a result of qualitative work will be supported in the relevant sections of the training. In the quantitative section of the research, the interactive web-assisted nurse program will take 1 week and the application will take 3 weeks. A text message will be sent to individuals to their phone to remind them to use the website. Messages will be sent twice a week, a total of 8 times. It will be used as Care Dependency, Body value, psychosocial Compliance to disease, website usability Scale measurement tools. After each assessment, the data obtained will be transferred to the "Social Sciences Software Statistical Package (SPSS).

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-75 who do not have communication problems,
* Patients who have undergone mastectomy for the first time,
* Patients who know their diagnosis,
* Patients with basic computer literacy,
* Patients with computer or internet access.
* Patients who agree to participate in the study will be included.

Exclusion Criteria:

* Patients with hearing, vision and understanding problems,
* Patients with metastases
* Patients with breast cyst excision,
* Patients with arm or shoulder limitation,
* Patients with breast reconstruction will not be included in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2022-08-24 (Actual); Primary Completion 2023-04-24 (Actual); Study Completion 2023-08-29 (Actual)

PRIMARY OUTCOMES:
Body Appreciation Scale | Before application
  It was developed in order to evaluate the extent to which individuals have positive thoughts about their own bodies and whether they respect these thoughts. Body Value Scale-2 is a 5-point Likert type measurement tool and consists of 10 items.There is no reverse item in the Body Value Scale and a minimum of 10 and a maximum of 50 points can be obtained from the scale. A total score is obtained by summing the scores of the items in the scale. A low score from the scale indicates that individuals have negative body values, while high scores indicate positive body values.
Care Dependency Scale | Before application
  The care dependency scale is a scale consisting of a total of 17 items, including activities of daily living, and graded with 5-point Likert-type scoring. Grading 1 = completely dependent, 5 = immediately, immediately / completely independent. The lowest score to be taken from the scale is 17 and the highest score is 85. A high scale score indicates that the patient is independent in meeting his/her self-care needs, while a low scale score indicates that patients are dependent on others to meet their care needs.
Psychosocial Adjustment to Illness-Self-Report Scale | Before application
  It measures the interaction of individuals with other individuals and institutions that make up the sociocultural environment.
  The scale consists of 46 items. The questions in the scale are divided into 7 areas of psychosocial adjustment to the disease.
  In the scale, four descriptive expressions were used to determine the varying levels of agreement for each question. The subject can choose the answer that best describes his or her personal experience. The items in the scale are given scores ranging from 0 to 3, and the answers are converted into numerical values. For each item in the scale, mostly negative changes since the disease are evaluated with 3 points, no change or positive changes are evaluated with 0 points. Low scores on the PAIS-SR scale indicate "good psychosocial adjustment" to the disease, and high scores indicate "poor psychosocial adjustment" to the disease. In the PAIS-SR, scores below 35 indicate "good psychosocial adjustment", scores between 35 and 51 indicate
Body Appreciation Scale | Immediately after application (1st week)
  It was developed in order to evaluate the extent to which individuals have positive thoughts about their own bodies and whether they respect these thoughts. Body Value Scale-2 is a 5-point Likert type measurement tool and consists of 10 items.There isno reverse item in the Body Value Scale and a minimum of 10 and a maximum of 50 points can be obtained from the scale. A total score is obtained by summing the scores of the items in the scale. A low score from the scale indicates that individuals have negative body values, while high scores indicate positive body values.
Care Dependency Scale | Immediately after application (1st week)
  The care dependency scale is a scale consisting of a total of 17 items, including activities of daily living, and graded with 5-point Likert-type scoring. Grading 1 = completely dependent, 5 = immediately, immediately / completely independent. The lowest score to be taken from the scale is 17 and the highest score is 85. A high scale score indicates that the patient is independent in meeting his/her self-care needs, while a low scale score indicates that patients are dependent on others to meet their care needs.
Psychosocial Adjustment to Illness-Self-Report Scale | Immediately after application (1st week)
  It measures the interaction of individuals with other individuals and institutions that make up the sociocultural environment.
Body Appreciation Scale | Immediately after application (3st week)
  It was developed in order to evaluate the extent to which individuals have positive thoughts about their own bodies and whether they respect these thoughts. Body Value Scale-2 is a 5-point Likert type measurement tool and consists of 10 items.
  There is no reverse item in the Body Value Scale and a minimum of 10 and a maximum of 50 points can be obtained from the scale. A total score is obtained by summing the scores of the items in the scale. A low score from the scale indicates that individuals have negative body values, while high scores indicate positive body values.
Care Dependency Scale | Immediately after application (3st week)
  The care dependency scale is a scale consisting of a total of 17 items, including activities of daily living, and graded with 5-point Likert-type scoring. Grading 1 = completely dependent, 5 = immediately, immediately / completely independent. The lowest score to be taken from the scale is 17 and the highest score is 85. A high scale score indicates that the patient is independent in meeting his/her self-care needs, while a low scale score indicates that patients are dependent on others to meet their care needs.
Psychosocial Adjustment to Illness-Self-Report Scale | Immediately after application (3st week)
  It measures the interaction of individuals with other individuals and institutions that make up the sociocultural environment.

SECONDARY OUTCOMES:
Website Usability Scale | Immediately after application
  The scale consists of a total of 25 questions with four sub-dimensions (ease of navigation = 10 questions, design = 7 questions, ease of access = 4 questions, ease of use = 4 questions). The answers to the items of the scale are collected with a Likert-type five-point rating scale. The scale consists of "Strongly agree (5)", "Agree (4)", "Undecided (3)", "Disagree (2)" and "Strongly disagree (1)". 21 of the items in the scale are positive and 4 of them are negative items. The lowest score to be taken from the scale is 25 and the highest score is 125.

CONTACTS AND LOCATIONS:
Overall Officials: Şeyda KAZANÇ, Lecturer, Principal Investigator — Cumhuriyet University; Şerife KARAGÖZOĞLU, Prof. Dr., Study Director — Cumhuriyet University
Locations (1):
- Gaziosmanpasa University, Tokat Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ab Malik N, Zhang J, Lam OL, Jin L, McGrath C. Effectiveness of computer-aided learning in oral health among patients and caregivers: a systematic review. J Am Med Inform Assoc. 2017 Jan;24(1):209-217. doi: 10.1093/jamia/ocw045. Epub 2016 Jun 6. PMID 27274013
- [Background] Adaylar M. Kronik hastalığı olan bireylerin hastalıktaki tutum, adaptasyon, algı ve öz-bakım yönelimleri. İstanbul Üniversitesi Sağlık Bilimleri Enstitüsü, Hemşirelik Anabilim Dalı, Doktora tezi, İstanbul, 1995
- [Background] Ahadzadeh AS, Sharif SP. Uncertainty and Quality of Life in Women With Breast Cancer: Moderating Role of Coping Styles. Cancer Nurs. 2018 Nov/Dec;41(6):484-490. doi: 10.1097/NCC.0000000000000552. PMID 29489477
- [Background] Anderson C, Islam JY, Elizabeth Hodgson M, Sabatino SA, Rodriguez JL, Lee CN, Sandler DP, Nichols HB. Long-Term Satisfaction and Body Image After Contralateral Prophylactic Mastectomy. Ann Surg Oncol. 2017 Jun;24(6):1499-1506. doi: 10.1245/s10434-016-5753-7. Epub 2017 Jan 5. PMID 28058563
- [Background] Akyolcu, N., Özhanlı Y., Kandemir D. (2019). Meme Kanserinde Güncel Gelişmeler. Sağlık Bilimleri ve Meslek Dergisi, 6(3), 583-94.
- [Background] Ayar, D., Öztürk, C. (2015). Tip 1 Diyabetik Ergenlerin Eğitiminde Yeni Yaklaşımlar Web Tabanlı Eğitim. Dokuz Eylül Üniversitesi Hemşirelik Fakültesi Elektronik Dergisi, 8 (3),184-189.
- [Background] Baysan Arabacı, L., Büyükbayram, A., Aktaş, Y., & Taşkın, N. (2018). Kronik ruhsal bozukluk tanısı alan hastaların bakım verenlerine verilen psikoeğitimin yaşadıkları güçlük ve psikososyal uyumlarına etkisi. Psikiyatri Hemşireliği Dergisi, 9(3), 175-185.
- [Background] Borosund E, Cvancarova M, Moore SM, Ekstedt M, Ruland CM. Comparing effects in regular practice of e-communication and Web-based self-management support among breast cancer patients: preliminary results from a randomized controlled trial. J Med Internet Res. 2014 Dec 18;16(12):e295. doi: 10.2196/jmir.3348. PMID 25525672
- [Background] Charnock D, Shepperd S, Needham G, Gann R. DISCERN: an instrument for judging the quality of written consumer health information on treatment choices. J Epidemiol Community Health. 1999 Feb;53(2):105-11. doi: 10.1136/jech.53.2.105. PMID 10396471
- [Background] Chow KM, So WKW, Choi KC, Chan CWH. Sexual function, psychosocial adjustment to illness, and quality of life among Chinese gynaecological cancer survivors. Psychooncology. 2018 Apr;27(4):1257-1263. doi: 10.1002/pon.4663. Epub 2018 Mar 1. PMID 29430767
- [Background] Classen CC, Chivers ML, Urowitz S, Barbera L, Wiljer D, O'Rinn S, Ferguson SE. Psychosexual distress in women with gynecologic cancer: a feasibility study of an online support group. Psychooncology. 2013 Apr;22(4):930-5. doi: 10.1002/pon.3058. Epub 2012 Feb 28. PMID 22374732
- [Background] Creswell, J. W., & Plano Clark, V. L. (2018). Designing and conducting mixed methods research. In (3 rd. ed.).
- [Background] Çakmak, E. K., Güneş, E., Çiftçi, S., & Üstündağ, M. T. (2011). Web Sitesi Kullan ı labilirlik Ölçe ğ inin Geli ş tirilmesi : Geçerlik , Güvenirlik Analizi ve Uygulama Sonuçlar ı Developing a Web Site Usability Scale : The Validity and Reliability Analysis & Implementation Results Giri ş. Pegem Eğitim ve Öğretim Dergisi, 1(2), 31-40.
- [Background] Çam, O., Saka, Ş., & Gümüş, A. B. (2009). Meme Kanserli Hastaların Psikososyal Uyumlarını Etkileyen Faktörlerin İncelenmesi. Meme Sagligi Dergisi/Journal of Breast Health, 5(2).
- [Background] Dauplat J, Kwiatkowski F, Rouanet P, Delay E, Clough K, Verhaeghe JL, Raoust I, Houvenaeghel G, Lemasurier P, Thivat E, Pomel C; STIC-RMI working group. Quality of life after mastectomy with or without immediate breast reconstruction. Br J Surg. 2017 Aug;104(9):1197-1206. doi: 10.1002/bjs.10537. Epub 2017 Apr 12. PMID 28401542
- [Background] Del Valle DD, Pardo JA, Maselli AM, Valero MG, Fan B, Seyidova N, James TA, Lee BT. Evaluation of online Spanish and English health materials for preventive mastectomy. are we providing adequate information? Breast Cancer Res Treat. 2021 May;187(1):1-9. doi: 10.1007/s10549-021-06171-1. Epub 2021 Mar 15. PMID 33721147
- [Background] Derogatis LR. The psychosocial adjustment to illness scale (PAIS). J Psychosom Res. 1986;30(1):77-91. doi: 10.1016/0022-3999(86)90069-3. PMID 3701670
- [Background] Dijkstra A, Sipsma D, Dassen T. Predictors of care dependency in Alzheimer's disease after a two-year period. Int J Nurs Stud. 1999 Dec;36(6):487-95. doi: 10.1016/s0020-7489(99)00044-9. PMID 10576119
- [Background] Diefenbach, M. A., Leventhal, H. (1996). The common-sense model of illness representation: Theoretical and practical considerations. Journal of Social Distress & the Homeless, 5(1): 11-38. https://doi.org/10.1007/BF02090456
- [Background] Dijkstra A, Kazimier H, Halfens RJ. Using the Care Dependency Scale for identifying patients at risk for pressure ulcer. J Adv Nurs. 2015 Nov;71(11):2529-39. doi: 10.1111/jan.12713. Epub 2015 Jun 23. PMID 26100573
- [Background] Doğu, Ö., Kaya, H., Gündüz, H., Parlak, S. (2015). Miyokard Enfarktüsü Geçirmiş Bireylere Eğitim ve Danışmanlıkta Web Tabanlı Uzaktan Eğitim Önerisi. MN Kardiyoloji, 22 (4):217-222. DOI: 10.2196/jmir.3749
- [Background] Elahi, N., Imanian, M., Zarea, K., Ahmadzadeh, A., & Karimyar Jahromi, M. (2017). Effect of continuous care model on body image among breast cancer patients undergoing chemotherapy: a clinical trial. International Journal of Cancer Management, 10(7).
- [Background] Elbaş, N. Ö. 2016. Cerrahi Hastalıkları Hemşireliği Akıl Notları, Meme hastalıkları cerrahisi ve hemşirelik bakımı. 1. Baskı. pp. 81-82. Ankara: Güneş Tıp Kitabevi
- [Background] Flitcroft K, Brennan M, Spillane A. Principles of patient-centred care and barriers to their implementation: a case study of breast reconstruction in Australia. Support Care Cancer. 2020 Apr;28(4):1963-1981. doi: 10.1007/s00520-019-04978-9. Epub 2019 Aug 2. PMID 31372747
- [Background] Gökdoğan F, Kır E, Özcan A, Cerit B, Yıldırım Y, Akbal S. Eğitim kitapçıkları güvenilir mi? 2. Uluslararası & IX. Ulusal Hemşirelik Kongresi Kongre Kitabı, Antalya, Türkiye, 2003:517-521.
- [Background] Gregorowitsch ML, van den Bongard HJGD, Young-Afat DA, Pignol JP, van Gils CH, May AM, Verkooijen HM. Severe depression more common in patients with ductal carcinoma in situ than early-stage invasive breast cancer patients. Breast Cancer Res Treat. 2018 Jan;167(1):205-213. doi: 10.1007/s10549-017-4495-y. Epub 2017 Sep 11. PMID 28894982
- [Background] Gu J, Groot G, Boden C, Busch A, Holtslander L, Lim H. Review of Factors Influencing Women's Choice of Mastectomy Versus Breast Conserving Therapy in Early Stage Breast Cancer: A Systematic Review. Clin Breast Cancer. 2018 Aug;18(4):e539-e554. doi: 10.1016/j.clbc.2017.12.013. Epub 2018 Jan 3. PMID 29396079
- [Background] Gutierrez Hermoso L, Velasco Furlong L, Sanchez-Roman S, Salas Costumero L. The Importance of Alexithymia in Post-surgery. Differences on Body Image and Psychological Adjustment in Breast Cancer Patients. Front Psychol. 2020 Dec 18;11:604004. doi: 10.3389/fpsyg.2020.604004. eCollection 2020. PMID 33391123
- [Background] Hawkins SD, Barilla S, Feldman SR. Web app based patient education in psoriasis - a randomized controlled trial. Dermatol Online J. 2017 Apr 15;23(4):13030/qt26d525z5. PMID 28541882
- [Background] Helms RL, O'Hea EL, Corso M. Body image issues in women with breast cancer. Psychol Health Med. 2008 May;13(3):313-25. doi: 10.1080/13548500701405509. PMID 18569899
- [Background] Ibrahim M, Muanza T, Smirnow N, Sateren W, Fournier B, Kavan P, Palumbo M, Dalfen R, Dalzell MA. Time course of upper limb function and return-to-work post-radiotherapy in young adults with breast cancer: a pilot randomized control trial on effects of targeted exercise program. J Cancer Surviv. 2017 Dec;11(6):791-799. doi: 10.1007/s11764-017-0617-0. Epub 2017 May 3. PMID 28470507
- [Background] Izydorczyk B, Kwapniewska A, Lizinczyk S, Sitnik-Warchulska K. Psychological Resilience as a Protective Factor for the Body Image in Post-Mastectomy Women with Breast Cancer. Int J Environ Res Public Health. 2018 Jun 5;15(6):1181. doi: 10.3390/ijerph15061181. PMID 29874874
- [Background] Jiao N, Zhu L, Chong YS, Chan WS, Luo N, Wang W, Hu R, Chan YH, He HG. Web-based versus home-based postnatal psychoeducational interventions for first-time mothers: A randomised controlled trial. Int J Nurs Stud. 2019 Nov;99:103385. doi: 10.1016/j.ijnurstu.2019.07.002. Epub 2019 Jul 21. PMID 31442783
- [Background] Kahissay MH, Fenta TG, Boon H. Beliefs and perception of ill-health causation: a socio-cultural qualitative study in rural North-Eastern Ethiopia. BMC Public Health. 2017 Jan 26;17(1):124. doi: 10.1186/s12889-017-4052-y. PMID 28122606
- [Background] Kankaya, B., Büyükaşık, S., Kapan, S., & Halil, A. (2019). Meme Kanseri Tedavisinde Güncel Yaklaşım/Current Management in Breast Cancer. Tıp Fakültesi Klinikleri Dergisi, 2(1), 7-10.
- [Background] Karakartal, D. (2018). Kanser Hastalarının Yaşadıkları Psiko-Sosyal Sorunların İncelenmesi. International Journal of Humanities and Education, 4(9), 48-62.
- [Background] Karamanoğlu, A. Y., & Özer, F. G. (2008). MASTEKTOMİLİ HASTALARDA EVDE BAKIM. Meme Sağlığı Dergisi, 4(1), 4-5.
- [Background] Kılıç, H. F., Cevheroğlu, S., & Görgülü, R. S. (2017). Dahiliye ve cerrahi kliniklerinde yatan hastaların bakım bağımlılığı düzeylerinin belirlenmesi. Dokuz Eylül Üniversitesi Hemşirelik Fakültesi Elektronik Dergisi, 10(1), 22-28.
- [Background] Kızıltan, G., Özaslan, C., Karaman, N., & Doğan, L. (2018). Early Wound Complications And Influencing Factors For The Breast Cancer Patients After Oncoplastic Surgery. AOT, 51(3), 416-423.
- [Background] Korkmaz S, Iyigun E, Tastan S. An Evaluation of the Influence of Web-Based Patient Education on the Anxiety and Life Quality of Patients Who Have Undergone Mammaplasty: a Randomized Controlled Study. J Cancer Educ. 2020 Oct;35(5):912-922. doi: 10.1007/s13187-019-01542-1. PMID 31119709
- [Background] Kugbey N, Oppong Asante K, Meyer-Weitz A. Illness perception and coping among women living with breast cancer in Ghana: an exploratory qualitative study. BMJ Open. 2020 Jul 14;10(7):e033019. doi: 10.1136/bmjopen-2019-033019. PMID 32665380
- [Background] Kuijpers W, Groen WG, Aaronson NK, van Harten WH. A systematic review of web-based interventions for patient empowerment and physical activity in chronic diseases: relevance for cancer survivors. J Med Internet Res. 2013 Feb 20;15(2):e37. doi: 10.2196/jmir.2281. PMID 23425685
- [Background] Eichhorn-Kissel J, Dassen T, Lohrmann C. Comparison of the responsiveness of the Care Dependency Scale for rehabilitation and the Barthel Index. Clin Rehabil. 2011 Aug;25(8):760-7. doi: 10.1177/0269215510397558. Epub 2011 Mar 14. PMID 21402648
- [Background] Korhan, E. A., Yönt, G. H., Tokem, Y., Karadağ, Ö., Sarıoğlu, E., & Yıldız, K. (2013). Dahİlİye Ve Cerrahİ Klİnİklerde Yatan Hastalarin Bakim Bağimliliği Düzeylerİnİn Belİrlenmesİ. Anadolu Hemşirelik ve Sağlık Bilimleri Dergisi, 16(4), 199-204.
- [Background] Kuntz S, Dassen T, Lahmann NA. Specific item patterns in comparison to generalized sum score-the Care Dependency Scale (CDS) as a screening tool for specific care problems. J Eval Clin Pract. 2018 Aug;24(4):731-739. doi: 10.1111/jep.12963. Epub 2018 Jun 8. PMID 29882621
- [Background] Kvillemo P, Branstrom R. Coping with breast cancer: a meta-analysis. PLoS One. 2014 Nov 25;9(11):e112733. doi: 10.1371/journal.pone.0112733. eCollection 2014. PMID 25423095
- [Background] Leventhal H, Phillips LA, Burns E. The Common-Sense Model of Self-Regulation (CSM): a dynamic framework for understanding illness self-management. J Behav Med. 2016 Dec;39(6):935-946. doi: 10.1007/s10865-016-9782-2. Epub 2016 Aug 11. PMID 27515801
- [Background] Mertens EI, Halfens RJ, Dietz E, Scheufele R, Dassen T. Pressure ulcer risk screening in hospitals and nursing homes with a general nursing assessment tool: evaluation of the care dependency scale. J Eval Clin Pract. 2008 Dec;14(6):1018-25. doi: 10.1111/j.1365-2753.2007.00935.x. Epub 2008 Feb 18. PMID 18284515
- [Background] Mike, S. (2018). Meme Kanseri Olan Kadınlarda Mastektomi Olanlar İle Mastektomi Olmayanların Depresyon Ve Umutsuzluk Düzeylerinin İncelenmesi (Master's thesis, İstanbul Gelişim Üniversitesi Sosyal Bilimler Enstitüsü).
- [Background] Mirandola D, Miccinesi G, Muraca MG, Sgambati E, Monaci M, Marini M. Evidence for adapted physical activity as an effective intervention for upper limb mobility and quality of life in breast cancer survivors. J Phys Act Health. 2014 May;11(4):814-22. doi: 10.1123/jpah.2012-0119. Epub 2013 Apr 5. PMID 23575310
- [Background] Moreira H, Canavarro MC. A longitudinal study about the body image and psychosocial adjustment of breast cancer patients during the course of the disease. Eur J Oncol Nurs. 2010 Sep;14(4):263-70. doi: 10.1016/j.ejon.2010.04.001. Epub 2010 May 21. PMID 20493769
- [Background] Nelson JA, Allen RJ Jr, Polanco T, Shamsunder M, Patel AR, McCarthy CM, Matros E, Dayan JH, Disa JJ, Cordeiro PG, Mehrara BJ, Pusic AL. Long-term Patient-reported Outcomes Following Postmastectomy Breast Reconstruction: An 8-year Examination of 3268 Patients. Ann Surg. 2019 Sep;270(3):473-483. doi: 10.1097/SLA.0000000000003467. PMID 31356276
- [Background] Oktan, V., & Saylan, E. (2020). Beden Değeri Ölçeği-2'nin (BDÖ-2) Türkçe Adaptasyonu: Geçerlik ve Güvenirlik Çalışması Adaptation of The Body Appreciation Scale-2 (BAS-2) to Turkish: A Validity and Reliability Study. Mersin Üniversitesi Eğitim Fakültesi Dergisi, 16(1), 94-103.
- [Background] Özkan Tuncay, F., & Kars Fertelli, T. (2020). Kronik Böbrek Yetmezliği Olan Bireylerde Bakım Bağımlılığı ve İlişkili Faktörler. Kocaeli Tıp Dergisi, 9(1), 32-40.
- [Background] Öztürkmen, A., Köroğlu, Ö., & Erkmen, H. (2019). Travma Sonrası Spinal Kord Hasarlı Bireylerin Sosyodemografik Özelliklerinin ve Psikososyal Uyumunun İncelenmesi. Journal of Physical Medicine & Rehabilitation Sciences/Fiziksel Tup ve Rehabilitasyon Bilimleri Dergisi, 22(3).
- [Background] Przezdziecki A, Sherman KA, Baillie A, Taylor A, Foley E, Stalgis-Bilinski K. My changed body: breast cancer, body image, distress and self-compassion. Psychooncology. 2013 Aug;22(8):1872-9. doi: 10.1002/pon.3230. Epub 2012 Dec 2. PMID 23203842
- [Background] Önal, D., Arabacı, L. B., & Mutlu, E. (2019). Miyokart infarktüsü geçiren hastalara bakım verenlerin bakım verme yükü ve psikososyal uyumları arasındaki ilişki. Turk J Cardiovasc Nurs, 10(23), 105-113.
- [Background] Puto G, Sowinska I, Scislo L, Walewska E, Kaminska A, Muszalik M. Sociodemographic Factors Affecting Older People's Care Dependency in Their Daily Living Environment According to Care Dependency Scale (CDS). Healthcare (Basel). 2021 Jan 21;9(2):114. doi: 10.3390/healthcare9020114. PMID 33494359
- [Background] Reigle BS, Wonders K. Breast cancer and the role of exercise in women. Methods Mol Biol. 2009;472:169-89. doi: 10.1007/978-1-60327-492-0_7. PMID 19107433
- [Background] Sağlık İstatistikleri Y (2015) https://www.saglikistatistikleri.gov. tr/dosyalar/SIY_ 2015.pdf. Erişim Tarihi: 25.05.2021.
- [Background] Shao J, Rodrigues M, Corter AL, Baxter NN. Multidisciplinary care of breast cancer patients: a scoping review of multidisciplinary styles, processes, and outcomes. Curr Oncol. 2019 Jun;26(3):e385-e397. doi: 10.3747/co.26.4713. Epub 2019 Jun 1. PMID 31285683
- [Background] Sivendran S, Jenkins S, Svetec S, Horst M, Newport K, Yost KJ, Yang M. Illness Understanding of Oncology Patients in a Community-Based Cancer Institute. J Oncol Pract. 2017 Sep;13(9):e800-e808. doi: 10.1200/JOP.2017.020982. Epub 2017 Jul 5. PMID 28678589
- [Background] Shah R, Al-Ajam Y, Stott D, Kang N. Obesity in mammaplasty: a study of complications following breast reduction. J Plast Reconstr Aesthet Surg. 2011 Apr;64(4):508-14. doi: 10.1016/j.bjps.2010.07.001. Epub 2010 Aug 3. PMID 20682461
- [Background] Toraman, S. (2021). Karma Yöntemler Araştırması: Kısa Tarihi, Tanımı, Bakış Açıları ve Temel Kavramlar. Nitel Sosyal Bilimler-Qualitative Social Sciences, 3(1), 1-29.
- [Background] Tosello G, Torloni MR, Mota BS, Neeman T, Riera R. Breast surgery for metastatic breast cancer. Cochrane Database Syst Rev. 2018 Mar 15;3(3):CD011276. doi: 10.1002/14651858.CD011276.pub2. PMID 29542106
- [Background] Turk KE, Yilmaz M. The Effect on Quality of Life and Body Image of Mastectomy Among Breast Cancer Survivors. Eur J Breast Health. 2018 Oct 1;14(4):205-210. doi: 10.5152/ejbh.2018.3875. eCollection 2018 Oct. PMID 30288494
- [Background] Tylka TL, Wood-Barcalow NL. The Body Appreciation Scale-2: item refinement and psychometric evaluation. Body Image. 2015 Jan;12:53-67. doi: 10.1016/j.bodyim.2014.09.006. Epub 2014 Oct 21. PMID 25462882
- [Background] Uğurlu, Z., & Akgün, H. S. (2019). Sağlık kurumlarına başvuran hastaların sağlık okuryazarlığının ve kullanılan eğitim materyallerinin sağlık okuryazarlığına uygunluğunun değerlendirilmesi. Mersin Univ Saglık Bilim Derg, 12(1), 96-106. https://doi.org/10.26559/mersinsbd.449973
- [Background] van Eck CF, Toor A, Banffy MB, Gambardella RA. Web-Based Education Prior to Outpatient Orthopaedic Surgery Enhances Early Patient Satisfaction Scores: A Prospective Randomized Controlled Study. Orthop J Sports Med. 2018 Jan 26;6(1):2325967117751418. doi: 10.1177/2325967117751418. eCollection 2018 Jan. PMID 29399589
- [Background] Varelas L, Egro FM, Evankovich N, Nguyen V. A Randomized Controlled Trial to Assess the Use of a Virtual Decisional Aid to Improve Knowledge and Patient Satisfaction in Women Considering Breast Reconstruction Following Mastectomy. Cureus. 2020 Dec 10;12(12):e12018. doi: 10.7759/cureus.12018. PMID 33457123
- [Background] Velasco L, Gutierrez Hermoso L, Alcocer Castillejos N, Quiroz Friedman P, Penacoba C, Catala P, Sanchez-Roman S. Association between quality of life and positive coping strategies in breast cancer patients. Women Health. 2020 Oct;60(9):1063-1069. doi: 10.1080/03630242.2020.1802398. Epub 2020 Aug 4. PMID 32752953
- [Background] Vuong B, Graff-Baker AN, Yanagisawa M, Chang SB, Mentakis M, Shim V, Knox M, Romero L, Kuehner G. Implementation of a Post-mastectomy Home Recovery Program in a Large, Integrated Health Care Delivery System. Ann Surg Oncol. 2019 Oct;26(10):3178-3184. doi: 10.1245/s10434-019-07551-0. Epub 2019 Aug 8. PMID 31396779
- [Background] Wan ES, Kantorowski A, Homsy D, Teylan M, Kadri R, Richardson CR, Gagnon DR, Garshick E, Moy ML. Promoting physical activity in COPD: Insights from a randomized trial of a web-based intervention and pedometer use. Respir Med. 2017 Sep;130:102-110. doi: 10.1016/j.rmed.2017.07.057. Epub 2017 Jul 25. PMID 29206627
- [Background] Wang TJ, Lu MH, Kuo PL, Chen YW, Lee SC, Liang SY. Influences of facial disfigurement and social support for psychosocial adjustment among patients with oral cancer in Taiwan: a cross-sectional study. BMJ Open. 2018 Nov 25;8(11):e023670. doi: 10.1136/bmjopen-2018-023670. PMID 30478118
- [Background] Weber WP, Soysal SD, El-Tamer M, Sacchini V, Knauer M, Tausch C, Hauser N, Gunthert A, Harder Y, Kappos EA, Schwab F, Fitzal F, Dubsky P, Bjelic-Radisic V, Reitsamer R, Koller R, Heil J, Hahn M, Blohmer JU, Hoffmann J, Solbach C, Heitmann C, Gerber B, Haug M, Kurzeder C. First international consensus conference on standardization of oncoplastic breast conserving surgery. Breast Cancer Res Treat. 2017 Aug;165(1):139-149. doi: 10.1007/s10549-017-4314-5. Epub 2017 Jun 3. PMID 28578506
- [Background] Wilson DJ. Exercise for the Patient after Breast Cancer Surgery. Semin Oncol Nurs. 2017 Feb;33(1):98-105. doi: 10.1016/j.soncn.2016.11.010. Epub 2017 Jan 4. PMID 28063632
- [Background] Wyatt KD, Jenkins SM, Plevak MF, Venegas Pont MR, Pruthi S. A personalized, web-based breast cancer decision making application: a pre-post survey. BMC Med Inform Decis Mak. 2019 Oct 21;19(1):196. doi: 10.1186/s12911-019-0924-7. PMID 31638964
- [Background] Yalçın, S., Arpa, Y., Cengiz, A., Doğan, S. 2015. Hemşirelerin hastaların taburculuk eğitim gereksinimlerine yönelik görüşleri ile hastaların eğitim gereksinimlerine yönelik görüşlerinin karşılaştırılması. Hemşirelikte Eğitim ve Araştırma Dergisi; 12 (3), 204-209
- [Background] Yi M, Kim J, Noh DY, Lee JL, Yoo KY, Hwang KT, Chung HD. Evaluation of the satisfaction and usefulness of a web-based educational program for breast cancer patients. Open Med Inform J. 2008;2:129-37. doi: 10.2174/1874431100802010129. Epub 2008 Aug 26. PMID 19415141
- [Background] Yönt, G. H., Akın, K. E., Khorshid, L., Eşer, İ., & Dijkstra, A. (2010). Bakım bağımlılığı ölçeğinin (Care Dependency Scale) yaşlı bireylerde geçerlik ve güvenirliğinin incelenmesi, Turkish Journal of Geriatrics Özel Sayı, 13: 71.
- [Background] Zhang P, Li CZ, Wu CT, Jiao GM, Yan F, Zhu HC, Zhang XP. Comparison of immediate breast reconstruction after mastectomy and mastectomy alone for breast cancer: A meta-analysis. Eur J Surg Oncol. 2017 Feb;43(2):285-293. doi: 10.1016/j.ejso.2016.07.006. Epub 2016 Jul 27. PMID 27503441
- [Background] Zeynep, Ş. E. N., Ersoy, A., Serel, S., Emiroğlu, M., Gülhan, S., & Soykan, A.(2018). Plastik ve Rekonstrüktif Cerrahi Girişimlerin Psikiyatrik Yönleri. Türk Plastik Rekonstrüktif Ve Estetik Cerrahi Dergisi, 11(2).